CLINICAL TRIAL: NCT03873402
Title: A Phase 3b, Randomized, Double-blind Study of Nivolumab Combined With Ipilimumab Versus Nivolumab Monotherapy for Patients With Previously Untreated Advanced Renal Cell Carcinoma and Intermediate- or Poor-Risk Factors
Brief Title: A Study of Nivolumab Combined With Ipilimumab Versus Nivolumab Alone in Participants With Advanced Kidney Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-8Y8; 2018-004695-35 (EudraCT Number)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + ipilimumab (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab + ipilimumab placebo (Experimental)
  Interventions: Other: Ipilimumab placebo

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Nivolumab + ipilimumab
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Nivolumab + ipilimumab
Other: Ipilimumab placebo — Specified dose on specified days
  Arms: Nivolumab + ipilimumab placebo

SUMMARY:
The purpose of this study is to test the effectiveness and safety of nivolumab combined with ipilimumab compared to nivolumab monotherapy in participants with previously untreated kidney cancer that has spread.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histological confirmation of renal carcinoma with clear cell component including participants who may have sarcomatoid features.
* Advanced (not amenable to curative surgery or radiation therapy) renal cell carcinoma (RCC) or metastatic RCC (mRCC).
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) criteria.
* No prior systemic therapy for RCC
* Must be intermediate or poor risk as per International Metastatic RCC Database Consortium (IMDC).

Exclusion Criteria:

* Any active central nervous system (CNS) metastases.
* Active, known, or suspected autoimmune disease.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody, or any other agents specifically targeting T-cell co-stimulation or checkpoint pathways

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2027-03-11 (Estimated); Study Completion 2027-03-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) by blinded independent central review (BICR) | Up to 34 months
Objective response rate (ORR) by BICR | Up to 23 months

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 4 years
Overall response rate (ORR) by investigator | Up to 4 years
Disease control rate (DCR) by investigator | Up to 4 years
Duration of response (DoR) by investigator | Up to 4 years
Time to objective response (TTR) by investigator | Up to 4 years
Progression Free Survival (PFS) by investigator | Up to 4 years
Progression free survival secondary objective (PFS2) by investigator | Up to 4 years
Disease control rate (DCR) by BICR | Up to 4 years
Duration of response (DoR) by BICR | Up to 4 years
Time to objective response (TTR) by BICR | Up to 4 years
Incidence of Adverse Events (AEs) | Up to 4 years
Incidence of drug-related AEs | Up to 4 years
Incidence of Severe Adverse Events (SAEs) | Up to 4 years
Incidence of drug-related SAEs | Up to 4 years
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 4 years
Incidence of clinically significant changes in clinical laboratory results: Coagulation tests | Up to 4 years
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 4 years
Incidence of clinically significant changes in clinical laboratory results: Serology tests | Up to 4 years
PFS based on gene expression (GEP) signatures | Up to 4 years
Objective response rate (ORR) based on GEP signatures | Up to 4 years
OS based on GEP signatures | Up to 4 years
OS based on programmed cell death protein ligand-1 (PD-L1) expression | Up to 4 years
ORR by BICR based on PD-L1 expression | Up to 4 years
PFS by BICR based on PD-L1 expression | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (78):
- United States (7):
  - Local Institution - 0013, Washington D.C., District of Columbia
  - Local Institution - 0053, Athens, Georgia
  - Local Institution - 0066, Boston, Massachusetts
  - Local Institution - 0088, Boston, Massachusetts
  - Local Institution - 0086, Boston, Massachusetts
  - The Reading Hosp Med Ctr Reg Cancer Ctr, West Reading, Pennsylvania
  - Local Institution - 0084, Charleston, South Carolina
- Argentina (7):
  - Local Institution - 0100, Capital Federal, Buenos Aires
  - Local Institution - 0011, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0060, Mar del Plata, Buenos Aires
  - Local Institution - 0025, Río Cuarto, Córdoba Province
  - Local Institution - 0001, Viedma, Río Negro Province
  - Local Institution - 0005, Córdoba
  - Local Institution - 0002, San Juan
- Austria (3):
  - Local Institution - 0033, Graz
  - Local Institution - 0031, Vienna
  - Local Institution - 0032, Wels
- Chile (5):
  - Local Institution - 0004, Viña del Mar, Región de Valparaíso
  - Local Institution - 0012, Viña El Mar, Región de Valparaíso
  - Local Institution - 0017, Independencia, Santiago Metropolitan
  - Local Institution - 0003, Santiago, Santiago Metropolitan
  - Local Institution - 0034, Santiago, Santiago Metropolitan
- Czechia (4):
  - Local Institution - 0020, Brno, South Moravian
  - Local Institution - 0097, Brno
  - Local Institution - 0019, Prague
  - Local Institution - 0018, Prague
- France (15):
  - Local Institution - 0096, Nice, Alpes-Maritimes
  - Local Institution - 0074, Brest, Finistère
  - Local Institution - 0078, Nancy, Meurthe-et-Moselle
  - Local Institution - 0091, Valenciennes, Nord
  - Local Institution - 0073, Angers
  - Local Institution - 0069, Angers
  - Local Institution - 0075, Besançon
  - Local Institution - 0094, Caen
  - Local Institution - 0081, Hyères
  - Local Institution - 0080, La Tronche
  - Local Institution - 0071, Marseille
  - Local Institution - 0092, Paris
  - Local Institution - 0093, Strasbourg
  - Local Institution - 0072, Suresnes
  - Local Institution - 0068, Villejuif
- Greece (2):
  - Local Institution - 0023, Athens
  - Local Institution - 0024, Larissa
- Italy (6):
  - Local Institution - 0082, Brescia, Lombardy
  - Local Institution - 0014, Arezzo
  - Local Institution - 0016, Aviano (PN)
  - Local Institution - 0021, Milan
  - Local Institution - 0015, Parma
  - Local Institution - 0077, Roma
- Mexico (6):
  - Local Institution - 0006, Mexico City, Mexico City
  - Local Institution - 0009, Mexico City, Mexico City
  - Local Institution - 0010, Mexico City, Mexico City
  - Local Institution - 0067, Monterrey, Nuevo León
  - Local Institution - 0008, Chihuahua City
  - Local Institution - 0046, Querétaro
- Poland (6):
  - Local Institution - 0030, Biała Podlaska
  - Local Institution - 0095, Bydgoszcz
  - Local Institution - 0062, Bytom
  - Local Institution - 0026, Gdansk
  - Local Institution - 0029, Poznan
  - Local Institution - 0027, Warsaw
- Local Institution - 0050, Lisbon, Portugal
- Romania (3):
  - Local Institution - 0061, Bucharest
  - Local Institution - 0056, Cluj-Napoca
  - Local Institution - 0065, Craiova
- Russia (2):
  - Local Institution - 0054, Saint Petersburg, Sankt-Peterburg
  - Local Institution - 0058, Novosibirsk
- Spain (11):
  - Local Institution - 0038, Barcelona
  - Local Institution - 0037, Barcelona
  - Local Institution - 0042, Córdoba
  - Local Institution - 0036, Madrid
  - Local Institution - 0035, Madrid
  - Local Institution - 0045, Pamplona
  - Local Institution - 0039, Sabadell
  - Local Institution - 0043, Santander
  - Local Institution - 0044, Santiago Compostela
  - Local Institution - 0041, Seville
  - Local Institution - 0040, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Individual patient level data from this study may be shared with qualified researchers, upon request, following the timelines and process detailed on https://www.bms.com/researchers-and-partners/independent-research/data-sharing-request-process.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03873402.html